CLINICAL TRIAL: NCT06967467
Title: Optimizing Antibiotic Selection in Hematologic Malignancy Patients With Reported Beta-lactam Allergy
Brief Title: Allergy Delabeling in Antibiotic Stewardship - Evaluations
Acronym: RENEW-EVAL
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Ebbing Lautenbach, Professor of Medicine and Epidemiology, University of Pennsylvania
Other Study IDs: 855769; R01HS029879 (AHRQ)
Record Dates: First submitted 2025-04-08; First posted 2025-05-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Beta Lactam Allergy in Patients With a Hematologic Malignancy
Keywords: penicillin allergy; hematologic cancer; allergy delabeling
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients who enroll in the RENEW intervention: Patients who agree to actively participate in the RENEW intervention designed to identify opportunities to have the beta lactam allergy label removed from their electronic medical record.
  Interventions: Behavioral: Semi-structured interview; Behavioral: Survey
- Patients who decline enrollment in the RENEW intervention: Patients who were approached for enrollment in the RENEW intervention but declined consent.
  Interventions: Behavioral: Semi-structured interview
- Clinicians: Clinicians who provide clinical care to patients enrolled in the intervention.
  Interventions: Behavioral: Survey; Behavioral: Semi-structured interview
- RENEW Clinical Pharmacist: The RENEW Clinical Pharmacist will screen, recruit, and consent potential participants and perform the RENEW intervention.
  Interventions: Behavioral: Ethnographic observation

INTERVENTIONS:
Behavioral: Semi-structured interview — Interviews designed to obtain information about patient reasons for enrolling or declining participation in the RENEW Intervention
  Groups: Patients who decline enrollment in the RENEW intervention; Patients who enroll in the RENEW intervention
Behavioral: Survey — Survey which will incorporate a series of closed-ended questions eliciting attitudes about the feasibility and acceptability of the intervention, allergy delabeling and future BL antibiotic use
  Groups: Patients who enroll in the RENEW intervention
Behavioral: Ethnographic observation — Observations designed to identify communication and contextual barriers to the implementation of RENEW
  Groups: RENEW Clinical Pharmacist
Behavioral: Survey — Survey instruments will measure knowledge,attitudes, and practices surrounding allergy delabeling and antibiotic stewardship in patients with HM and perceptions of the feasibility and acceptability of the RENEW intervention
  Groups: Clinicians
Behavioral: Semi-structured interview — Interviews designed to obtain information from clinicians about their perception of the implementation of the RENEW intervention
  Groups: Clinicians

SUMMARY:
The goal of this RENEW-EVAL project is to understand the potential barriers to implementation of the RENEW intervention into the routine clinical care of patients with a hematological malignancy.

DETAILED DESCRIPTION:
The RENEW clinical intervention is designed to evaluate the impact of a comprehensive beta lactam (BL) allergy delabeling intervention on clinical outcomes among patients hospitalized with a hematologic malignancy (HM). HM patients are at a high risk of infection-related complications but are limited to antibiotic therapy based on self-reported allergies. The RENEW intervention will test the impact of a pharmacist-led BL allergy delabeling intervention on clinical outcomes and antibiotic use in hospitalized patients with HM.

The implementation of clinical interventions are often affected by non-clinical factors including workflow challenges and the beliefs of patients, their families, and clinical staff.

The RENEW-EVAL study is a concurrent mixed methods process evaluation of the RENEW intervention that aims to identify the social and behavioral factors that shape implementation of the intervention and to measure implementation outcomes including feasibility, acceptability, and fidelity.

Three types of data will be gathered by the research team as part of the RENEW-EVAL project: 1) semistructured interviews with patients and clinicians, (2) ethnographic observations of the delivery of the RENEW intervention, and 3) surveys assessing patient and clinician attitudes towards BL allergy delabeling, and implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patient participants:

* a diagnosis of a hematologic malignancy (lymphoma, leukemia, myeloma)
* a prior label applied to their medical record to indicate a beta lactam allergy
* hospitalized as an inpatient to an oncology service at the time the study is conducted

Clinician participants:

* member of the primary inpatient care team

Exclusion Criteria:

Patient participants:

* meet one of the exclusionary criteria for the RENEW clinical intervention

Clinician participants:

* no exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patient participants who are admitted to an inpatient oncology service at the Hospital of the University of Pennsylvania, and clinician participants who provide clinical care during the admission. By definition, the Clinical Pharmacist who enrolls patient participants will also be part of the study population.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Implementation | From baseline Month 1 to Month 36
  Feasibility of implementation among clinicians and patients measured by questionnaire. Items are adapted from the validated Feasibility of Implementation Measure (FIM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better feasibility. The items are analyzed individually and not summed to a total score.
Acceptability of Implementation | From baseline Month 1 to Month 36
  Acceptability of implementation among clinicians and patients measured by questionnaire. Items are adapted from the validated Acceptability of Implementation Measure (AIM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better acceptability. The items are analyzed individually and not summed to a total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States